CLINICAL TRIAL: NCT02711943
Title: Non-interventional (Observational) Study of the Administration of Levolet® R, Film-coated Tablets (Dr. Reddy's Laboratories Ltd., India) in Adults With Chronic Prostatitis in Routine Clinical Practice
Brief Title: Non Interventional Study of Levofloxacin in Chronic Prostatitis
Acronym: Levolet-R
Status: Completed | Type: Observational
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: DRL_RUS/MD/2013/PMS/LEVOLET R
Record Dates: First submitted 2016-03-14; First posted 2016-03-17 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Chronic Prostatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Levofloxacin 500 — Oral levofloxacin (Levolet®) at a dose of 500 mg once a day for 28 days
  Other Names: Levolet R

SUMMARY:
Chronic prostatitis is a common disease in men with the following typical symptoms decreasing the ability to work and quality of life: pain, urination disorders, copulatory dysfunction.

Following study is conducted to study Levofloxacin in chronic prostatitis.

DETAILED DESCRIPTION:
Chronic prostatitis is a common disease in men with the following typical symptoms decreasing the ability to work and quality of life: pain, urination disorders, copulatory dysfunction. Professional societies recommend diagnosing and treating patients with chronic prostatitis on the basis of determination of belonging to classification categories proposed by the National Institute of Diabetes and Digestive and Kidney Diseases and the National Institutes of Health in the USA .

According to the recommendations of European Association of Urologists, in chronic bacterial inflammation of the prostate and in nonbacterial (inflammatory syndrome of chronic pelvis pain), the performance of antibacterial therapy during four - six weeks is efficient. The first-line drugs are fluoroquinolones (ciprofloxacin and levofloxacin) as along with good tolerance they easily penetrate into the zones of the prostate inflammation and are highly efficient in respect of prostatitis pathogens . Although the treatment with levofloxacin promotes more evident decrease in clinical symptoms and demonstrates better parameters of eradication of pathogen in comparison with ciprofloxacin administration, it is used less common, possibly due to insufficient awareness of physicians of its high efficacy in chronic prostatitis .

ELIGIBILITY:
Inclusion Criteria:

* male patients aged from 18 to 60 years, inclusive, with a diagnosis of the chronic prostatitis, which appointed the drug Levolet® P as a causal treatment.
* Demonstrated sensitivity to levofloxacin abjection of chronic bacterial prostatitis.
* The presence of a written informed consent to participate in research

Exclusion Criteria:

* participation in another clinical study during the period of this study.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with chronic prostatitis, age 18-60 years
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2013-07; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with response as per IMPSS scale | 28 days
  Subjective evaluation of the treatment was performed using Integrative Medicine Patient Satisfaction Scale - IMPSS: completely satisfied, satisfied, neutral attitude, unsatisfied and extremely unsatisfied.

SECONDARY OUTCOMES:
Percentage of patients response as per IMOS | 28 days
  Therapy results were evaluated using physician's opinion according to Integrative Medicine Outcome Scale - IMOS (complete recovery, significant improvement, insignificant to moderate improvement, no changes, deterioration)

CONTACTS AND LOCATIONS:
Overall Officials: IGOR A KORNEYEV, Principal Investigator — Acad. I.P. Pavlov First Saint-Petersburg State Medical University

IPD SHARING:
Plan to Share IPD: No